CLINICAL TRIAL: NCT03221127
Title: Kuopio Ischaemic Heart Disease Risk Factor Study (Nutrition Component)
Status: Active, not recruiting | Type: Observational
Sponsor: University of Eastern Finland (Other)
Responsible Party: Sponsor
Other Study IDs: KIHD Nutrition
Record Dates: First submitted 2017-07-07; First posted 2017-07-18 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Cardiovascular Diseases; Diabetes; Metabolic Syndrome; Cancer; Inflammatory Disease; Atherosclerosis; Cognitive Decline; Liver Diseases; Death; Pain, Chronic; Depression; Infection; Chronic Disease
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Metabolic Syndrome; Neoplasms; Atherosclerosis; Cognitive Dysfunction; Liver Diseases; Death; Chronic Pain; Depression; Infections; Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, serum, plasma, urine, hair, nails, DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To determine associations between dietary factors and risk of major chronic diseases and their risk factors

DETAILED DESCRIPTION:
STUDY POPULATION The Kuopio Ischaemic Heart Disease Risk Factor Study (KIHD) is an on-going prospective, population-based cohort study of risk factors for cardiovascular diseases, other chronic diseases and metabolic conditions in a sample of men from eastern Finland. The baseline examinations were carried out between 1984 and 1989, when 2,682 men (82.9% of those eligible) who were 42, 48, 54 or 60 years old were recruited. The first cohort consisted of 1166 men who were 54 years old, enrolled in 1984-1986, and the second cohort included 1516 men who were 42, 48, 54 or 60 years old, enrolled in 1986-1989. The baseline examinations were followed by the 4-year examinations (1991-1993), in which 1038 men from the second cohort (88% of the eligible) participated. At the 11-year examinations (1998-2001), all men from the second cohort were invited and 854 men (95% of the eligible) participated. These examinations were also the baseline for 920 postmenopausal women (78.4% of the 1173 eligible women) from the same area, aged 53-73 years. During the 20-year examination round, all men from the first and second baseline cohorts and all women were invited to the study site, and a total of 1241 men (80% of the eligible) and 634 women (81.0%) participated.

ASSESSMENT OF DIETARY INTAKES Food consumption has been assessed with an instructed food recording of four days, one of which was a weekend day, by household measures. A picture book of common foods and dishes was used to help in estimation of portion sizes. For each food item the participant could choose from 3-5 commonly used portion sizes or describe the portion size in relation to those in the book. In order to further improve accuracy, instructions were given and completed food records were checked by a nutritionist together with a participant. Nutrient intakes were estimated using the NUTRICA® 2.5 software (Social Insurance Institution, Turku, Finland). The databank of the software is mainly based on Finnish values of nutrient composition of foods.

OUTCOME ASSESSMENT Registration of the incidence of major chronic diseases and deaths during the follow up is based on the national registries (Hospital discharge registry, Cause of death register, Social Insurance Institution of Finland register for reimbursement of medicine expenses) by use of the Finnish personal identification code (social security number), and/or on findings at the re-examination rounds (such as fasting plasma glucose or 2-h oral glucose tolerance test to define type 2 diabetes in addition to data from the national registries).

ELIGIBILITY:
Inclusion Criteria:

* Aged 42, 48, 54 or 60 years (men at baseline in 1984-1989)
* Aged 53 to 73 years (women at their baseline in 1998-2001)
* Living in the city of Kuopio or neighboring rural areas

Exclusion Criteria:

* Condition that prevented visit at study clinic

Ages: 42 Years to 73 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: See "Detailed description"
Sampling Method: Probability Sample
Enrollment: 2682 (Actual)
Dates: Start 1984-03-01 (Actual); Primary Completion 2052-12-31 (Estimated); Study Completion 2052-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular disease | Annually between March 1984 and December 2052
  Incidence of cardiovascular disease
Carotid atherosclerosis | From baseline to 4-y, 11-y and 20-y examinations
  Progression of common carotid artery - intima-media thickness (CCA-IMT)
Death | Annually between March 1984 and December 2052
  Incidence of death

SECONDARY OUTCOMES:
Type 2 diabetes | Annually between March 1984 and December 2052
  Incidence of type 2 diabetes
Dementia | Annually between March 1984 and December 2052
  Incidence of dementia
Cancer | Annually between March 1984 and December 2052
  Incidence of cancer
Infectious disease | Annually between March 1984 and December 2052
  Incidence of hospitalization due infectious disease

CONTACTS AND LOCATIONS:
Overall Officials: Jussi Kauhanen, MD, PhD, Principal Investigator — University of Eastern Finland, Institute of Public Health and Clinical Nutrition

IPD SHARING:
Plan to Share IPD: Yes
Data available for collaborative projects

REFERENCES:
- [Derived] Hockey M, Hoare E, Mohebbi M, Tolmunen T, Hantunen S, Tuomainen TP, Macpherson H, Staudacher H, Jacka FN, Virtanen JK, Rocks T, Ruusunen A. Nonfermented Dairy Intake, but Not Fermented Dairy Intake, Associated with a Higher Risk of Depression in Middle-Age and Older Finnish Men. J Nutr. 2022 Aug 9;152(8):1916-1926. doi: 10.1093/jn/nxac128. PMID 35652820
- [Derived] Ylilauri MPT, Voutilainen S, Lonnroos E, Virtanen HEK, Tuomainen TP, Salonen JT, Virtanen JK. Associations of dietary choline intake with risk of incident dementia and with cognitive performance: the Kuopio Ischaemic Heart Disease Risk Factor Study. Am J Clin Nutr. 2019 Dec 1;110(6):1416-1423. doi: 10.1093/ajcn/nqz148. PMID 31360988
- [Derived] Abdollahi AM, Virtanen HEK, Voutilainen S, Kurl S, Tuomainen TP, Salonen JT, Virtanen JK. Egg consumption, cholesterol intake, and risk of incident stroke in men: the Kuopio Ischaemic Heart Disease Risk Factor Study. Am J Clin Nutr. 2019 Jul 1;110(1):169-176. doi: 10.1093/ajcn/nqz066. PMID 31095282
- [Derived] Virtanen HEK, Voutilainen S, Koskinen TT, Mursu J, Kokko P, Ylilauri MPT, Tuomainen TP, Salonen JT, Virtanen JK. Dietary proteins and protein sources and risk of death: the Kuopio Ischaemic Heart Disease Risk Factor Study. Am J Clin Nutr. 2019 May 1;109(5):1462-1471. doi: 10.1093/ajcn/nqz025. PMID 30968137
- [Derived] Virtanen HEK, Voutilainen S, Koskinen TT, Mursu J, Tuomainen TP, Virtanen JK. Intake of Different Dietary Proteins and Risk of Heart Failure in Men: The Kuopio Ischaemic Heart Disease Risk Factor Study. Circ Heart Fail. 2018 Jun;11(6):e004531. doi: 10.1161/CIRCHEARTFAILURE.117.004531. PMID 29844244
- See also: KIHD description and timeline — https://www.uef.fi/web/nutritionepidemiologists/kuopio-ischaemic-heart-disease-risk-factor-study-kihd-1984-